CLINICAL TRIAL: NCT03482687
Title: It's Your Game: An Innovative Approach to Preventing Teen Dating Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Melissa Peskin, Associate Professor, Department of Health Promotion and Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-12-0593
Record Dates: First submitted 2016-05-25; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Adolescent Behavior; Interpersonal Relationships; Domestic Violence; Physical Violence
Keywords: adolescent behavior; interpersonal relationships; intimate partner violence; violence/prevention & control; program evaluation; teen dating violence
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Me & You: Building Healthy Relationships (Experimental): Me & You: Building Healthy Relationships is a classroom- and computer-based healthy relationships curriculum for middle school students. It consists of thirteen 25-minute lessons: 5 classroom, 5 computer-only, and 3 classroom-computer hybrid.
  Interventions: Behavioral: Me & You: Building Healthy Relationships
- Comparison Group (No Intervention): No intervention was provided, only usual care.

INTERVENTIONS:
Behavioral: Me & You: Building Healthy Relationships — Me & You: Building Healthy Relationships is a classroom- and computer-based healthy relationships curriculum for middle school students. It consists of thirteen 25-minute lessons: 5 classroom, 5 computer-only, and 3 classroom-computer hybrid. The curriculum integrates group-based classroom activities (e.g., role-plays, group discussion, and other skill-building activities) and computer-based activities, some of which are individually tailored. The curriculum was adapted from an existing effective sex education and relationship curriculum, It's Your Game…Keep it Real (IYG), which was enhanced to more explicitly address teen dating violence (TDV).
  Arms: Me & You: Building Healthy Relationships

SUMMARY:
The purpose of this study is to evaluate Me & You: Building Healthy Relationships, a classroom- and computer-based healthy relationships and dating violence prevention curriculum for 6th grade students, in a large, urban public school district in Southeast Texas.

DETAILED DESCRIPTION:
The purpose of this three year study is to evaluate Me & You: Building Healthy Relationships, a classroom- and computer-based healthy relationships and dating violence prevention curriculum for 6th grade students, in a large, urban public school district in Southeast Texas. This curriculum was adapted from an existing effective sex education and relationship curriculum, It's Your Game…Keep it Real (IYG), which was enhanced to more explicitly address teen dating violence (TDV) and encompass multiple levels of the social-ecological model (e.g., youth, family, school staff). A randomized two-arm, nested design was conducted among 6th grade students, where students receiving the curriculum were compared to students receiving usual care. Ten middle schools participated in the study, five schools were randomly assigned to receive the curriculum and five to receive usual care. Outcomes were assessed at baseline, immediately following the intervention, and 12 months after baseline. Parental permission and student assent were obtained prior to administration of the surveys. The primary hypothesis is that students who receive the curriculum will have significantly lower TDV perpetration than those who do not receive the curriculum.

ELIGIBILITY:
Inclusion Criteria:

* 6th graders attending regular classes in ten study schools in large, urban school district in Southeast Texas

Exclusion Criteria:

* No students were excluded based on race/ethnicity, age, or gender.
* Students were informed that surveys and the intervention were only available in English and were asked to consider their comfort level with participating in the study.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 834 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent of youth who perpetrated any type of teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who were victimized by any type of teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.

SECONDARY OUTCOMES:
Percent of youth who perpetrated psychological teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who were victimized by psychological teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who perpetrated physical teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who were victimized by physical teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who perpetrated sexual teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who were victimized by sexual teen dating violence as indicated by the Conflict in Adolescent Dating Relationships Inventory | One year
  Validated self report measure by Wolfe et al.
Percent of youth who perpetrated electronic teen dating violence as indicated measures adapted from Picard and Zweig | One year
  Validated self report measure by Picard et al. and Zweig et al.
Percent of youth who were victimized by electronic teen dating violence as indicated measures adapted from Picard and Zweig | One year
  Validated self report measure by Picard et al. and Zweig et al.
Mean score reflecting student norms toward violence for boys and girls as indicated byt the Acceptance of Dating Abuse Survey | One year
  Validated self report measure by Foshee et al.
Mean score for self-efficacy to resolve conflict as indicated by the Teen Conflict Survey | One year
  Validated self report measure by Dahlberg et al.
Percent of youth reported one or more positive coping strategies as indicated by the Kidcope-Child Survey Form | One year
  Kidcope-Child Form by Laslo et al.
Mean score of constructive and destructive conflict resolution skills as indicated by valid scales developed by Foshee et al. | One year
  Validated self report measure by Foshee et al.
Mean score for attitudes towards sexting as indicated by a scale developed by Strassberg et al. | One year
  Validated self report measure by Strassberg et al.
Mean score related to a student's belief in the need for help for dating violence victimization as indicated by measures developed by Foshee et al. | One year
  Validated self report measure by Foshee et al.
Mean score for perceived peer dating violence perpetration (from the perspective of student) - newly developed | One year
  newly developed self-report measure
Mean score for parental communication about drugs, sex, and relationships as indicated by measures developed by Tharp et al. | One year
  Validated self report measure by Tharp and Noonan
Percent of youth who indicated social support from source as indicated by measures adapted from the Social Support Rating Scale | One year
  Validated self report measure by Cauce et al.
Percent of youth who perpetrated bullying as indicated by measures developed by Wang et al. | One year
  Validated self report measure by Wang et al.
Percent of youth who were victimized by bullying as indicated by measures developed from Wang et al. | One year
  Validated self report measure by Wang et al.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Peskin, PhD, Principal Investigator — University of Texas Houston School of Public Health; Susan Tortolero Emery, PhD, Principal Investigator — University of Texas Houston School of Public Health
Locations (1):
- Melissa Fleschler Peskin, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No